CLINICAL TRIAL: NCT03479073
Title: The Characteristics of Patients Experiencing Stroke or Systemic Embolism During Follow up Period After Atrial Fibrillation Ablation
Brief Title: Risk Factors of Stroke or Systemic Embolism After Atrial Fibrillation Ablation
Status: Completed | Type: Observational
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Principal Investigator, Hong Euy Lim, MD, Professor, Korea University Guro Hospital
Other Study IDs: KUGH17098-001
Record Dates: First submitted 2018-03-06; First posted 2018-03-27 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke group: Patients who experienced stroke or systemic embolic event following catheter ablation for AF.
- Control group: Patients who did not experienced stroke or systemic embolic event following catheter ablation for AF.

SUMMARY:
To investigate the rate and risk factors of stroke or systemic embolism (SE) following atrial fibrillation (AF) ablation.

DETAILED DESCRIPTION:
Since catheter ablation for AF reduces the burden of AF effectively, several studies have demonstrated that catheter ablation not only improves the quality of life but also reduces the risk of stroke and all cause mortality. However, until now the guideline has recommended the continuation of oral anticoagulation (OAC) therapy in patients who are at risk of stroke or systemic embolism (SE) based on the CHA2DS2-VASc score, even though they have sinus rhythm following catheter ablation. The aims of this retrospective study is to assess the rate of stroke/SE during follow-up period after AF ablation and identify the independent risk factors for stroke/SE in patients who underwent catheter ablation for AF.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent catheter ablation for AF

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population was extracted from a consortium of registry of AF ablation by three University Hospitals (Korea univ Guro, Korea univ Anam and Seoul National University) from 1998 to 2016.
Sampling Method: Non-Probability Sample
Enrollment: 3198 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2018-06-14 (Actual)

PRIMARY OUTCOMES:
Incidence of stroke or systemic embolism after AF ablation | From the time of catheter ablation until the date of the last visit or the date of event.(Retrospective period of up to 20 years)
  Risk factors for stroke or systemic embolism after AF ablation

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul National University Hospital, Seoul

REFERENCES:
- [Derived] Ahn J, Shin SY, Shim J, Kim YH, Han SJ, Choi EK, Oh S, Shin JY, Choe JC, Park JS, Lee HW, Oh JH, Choi JH, Lee HC, Cha KS, Hong TJ, Lip GYH, Lim HE. Association between epicardial adipose tissue and embolic stroke after catheter ablation of atrial fibrillation. J Cardiovasc Electrophysiol. 2019 Nov;30(11):2209-2216. doi: 10.1111/jce.14154. Epub 2019 Sep 19. PMID 31502330